CLINICAL TRIAL: NCT04950270
Title: The Arginine Vasopressin aXis as a Potential Therapeutic Target for Posterior REverSible Encephalopathy SyndromE (XPRESSE)
Brief Title: Copeptin Kinetics in Critically Ill Patients With Posterior Reversible Encephalopathy Syndrome
Acronym: XPRESSE
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH3-AOJCE20-BL-XPRESSE
Record Dates: First submitted 2021-06-14; First posted 2021-07-06 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Posterior Reversible Encephalopathy Syndrome
Keywords: Posterior Leukoencephalopathy Syndrome; Antidiuretic hormone; Intensive Care
MeSH Terms: conditions — Posterior Leukoencephalopathy Syndrome; Diabetes Insipidus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group: Critically ill adult patients meeting all eligibility criteria with MRI-based PRES diagnosis within the last 48 hours
  Interventions: Biological: Blood copeptin monitoring; Other: phone interview

INTERVENTIONS:
Biological: Blood copeptin monitoring — Blood copeptin monitoring during the first 6 days of ICU stay with PRES
Other: phone interview — Structured phone interview at 3 months to collect vital status and modified Rankin Scale score

SUMMARY:
XPRESSE is a multicenter observational prospective biomarker study in which critically ill patients with MRI-based PRES diagnosis will have copeptin kinetics from a daily blood sample for 6 days and a 3-month follow-up. This study aims to investigate the relationship between copeptin and PRES in order to establish the optimal therapeutic time window for vaptan treatment against PRES.

Data collection using an electronic case report form will include demographic data, medical history and data related to PRES: onset modalities and date of symptoms control, radiological features of PRES, biological investigations, results of etiological investigations and therapeutic management (e.g., anticonvulsants, antihypertensive drugs, supportive treatments). Outcomes will include modified Rankin scale score and Glasgow Outcome Scale score at ICU discharge, 3-month modified Rankin Scale score and 3-month mortality.

DETAILED DESCRIPTION:
Posterior reversible encephalopathy syndrome (PRES) is a clinical and radiological entity associating various neurological manifestations (e.g., encephalopathy, seizures) with a typical subcortical brain edema. While the pathophysiology of PRES remains elusive, the involvement of the arginine vasopressin (AVP) axis has recently been suggested by its stimulation in almost all etiologies of PRES as well as by its pathogenesis in the generation of brain edema that has been established in different preclinical models (e.g., traumatic brain injury, intracerebral hemorrhage) (Largeau et al., Mol Neurobiol 2019 - PMID: 30924075). Copeptin, a stable peptide derived from the same precursor as AVP and released in an equimolar ratio to AVP, is largely used in vivo to monitor AVP secretion. In a series of 225 critically ill patients free from PRES, median copeptin admission level was 50 pmol/L (Krychtiuk et al., PLOS ONE 2017- PMID: 28118414). By analogy to copeptin kinetics in patients with traumatic brain injury (Dong et al., J Trauma 2011 - PMID: 21502880), copeptin could attain peak level during the first week of PRES.

Blocking vasopressin receptors with vaptan appears to be a promising approach for PRES treatment. This study aims to investigate the relationship between copeptin and PRES in order to establish the optimal therapeutic time window for vaptan treatment against PRES.

XPRESSE is a multicenter observational prospective biomarker study in which critically ill patients in 4 French ICUs with MRI-based PRES diagnosis will have copeptin kinetics from a daily blood sample for 6 days and a 3-month follow-up.

Data collection using an eCRF will include demographic data, medical history and data related to PRES: onset modalities and date of symptoms control, radiological features of PRES, biological investigations, results of etiological investigations and therapeutic management (e.g., anticonvulsants, antihypertensive drugs, supportive treatments). Outcomes will include modified Rankin scale score and Glasgow Outcome Scale score at ICU discharge, 3-month modified Rankin Scale score and 3-month mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years ;
* Obtaining the non-opposition ;
* Patient hospitalized in ICU;
* PRES diagnosed within the last 48 hours (before admission or during ICU stay), based on the following clinico-radiological criteria :

  * Presentation with acute clinical symptoms ;
  * Presence of known risk factor for PRES;
  * Distributions of T2 weighted imaging (T2WI) or T2-fluid attenuated inversion recovery (T2-FLAIR) hyperintensities compatible with PRES imaging patterns ;
  * No other possible causes of these neuroimaging abnormalities found.

Exclusion Criteria:

* Patient under legal protection ;
* Patient under guardianship or curatorship
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill adult patients in ICU with PRES
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2022-06-18 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-02-26 (Actual)

PRIMARY OUTCOMES:
Estimation of time to maximum blood copeptin concentration (Tmax) | Up to 120 hours post-baseline
  Tmax will be estimated from copeptin kinetics: 6 samples at about 24 hours interval during the first 6 days of ICU stay with PRES

SECONDARY OUTCOMES:
Estimation of Tmax according to the etiology of PRES | Up to 120 hours post-baseline
Estimation of Tmax according to the type of MRI-based brain edema at diagnosis | Up to 120 hours post-baseline
  Diffusion-weighted imaging (DWI) sequences and Apparent diffusion coefficient (ADC) maps will be used to discriminate a cytotoxic pattern of edema from a vasogenic edema
Estimation of Area Under the Curve from D0 to D5 (AUC D0-D5) of blood copeptin according to the etiology of PRES | Up to 120 hours post-baseline
  AUC D0-D5 will be estimated from copeptin kinetics: 6 samples at about 24 hours interval during the first 6 days of ICU stay with PRES
Estimation of AUC D0-D5 of blood copeptin according to the type of MRI-based brain edema at diagnosis | Up to 120 hours post-baseline
  DWI sequences and ADC maps will be used to discriminate a cytotoxic pattern of edema from a vasogenic edema
Estimation of time to reach a copeptin concentration ≤50 pmol/L according to the etiology of PRES | Up to 120 hours post-baseline
Estimation of time to reach a copeptin concentration ≤50 pmol/L according to the type of MRI-based brain edema at diagnosis | Up to 120 hours post-baseline
  DWI sequences and ADC maps will be used to discriminate a cytotoxic pattern of edema from a vasogenic edema
Correlation analysis between AUC D0-D5 of blood copeptin and the extent of T2-FLAIR hyperintensities at diagnosis | Up to 120 hours post-baseline
Correlation analysis between AUC D0-D5 of blood copeptin and ADC values at diagnosis | Up to 120 hours post-baseline
Association analysis between AUC D0-D5 of blood copeptin and cerebral hemorrhagic lesions at diagnosis | Up to 120 hours post-baseline
Association analysis between AUC D0-D5 of blood copeptin and contrast enhancement in the brain at diagnosis | Up to 120 hours post-baseline
Correlation analysis between AUC D0-D5 of blood copeptin and AUC D0-D5 of mean arterial pressure | Up to 120 hours post-baseline
Correlation analysis between AUC D0-D5 of blood copeptin and AUC D0-D5 of serum creatinine | Up to 120 hours post-baseline
Association analysis between AUC D0-D5 of blood copeptin and Glasgow Outcome Scale score < 4 at ICU discharge | 0, 24, 48, 72, 96, 120 hours post-baseline and ICU discharge
  Glasgow Outcome Scale score: [1: Death, 2: Persistent vegetative state, 3: Severe disability, 4: Moderate disability, 5: Low disability]
Association analysis between AUC D0-D5 of blood copeptin and modified Rankin Scale score ≥ 4 at 3-month follow-up | 0, 24, 48, 72, 96, 120 hours post-baseline and 3 months
  Day-90 modified Rankin scale will be determined during a structured phone interview.
  Modified Rankin Scale score: [0: No symptoms at all, 1: No significant disability, 2: Slight disability, 3: Moderate disability, 4: Moderately severe disability, 5: Severe disability]
Association analysis between AUC D0-D5 of blood copeptin and mortality at 3-month follow-up | 0, 24, 48, 72, 96, 120 hours post-baseline and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Bérenger LARGEAU, PharmD, Study Chair — University Hospital, Tours; Charlotte SALMON GANDONNIERE, MD, PhD, Principal Investigator — University Hospital, Tours
Locations (4):
- France (4):
  - University hospital, Nantes
  - Hospital, Orléans
  - University hospital, Rennes
  - University hospital, Tours

IPD SHARING:
Plan to Share IPD: Undecided